CLINICAL TRIAL: NCT01404065
Title: Investigation of the Mechanisms of Transcranial Direct Current Stimulation of Motor Cortex Coupled With Visual Illusion for the Treatment of Chronic Pain in Spinal Cord Injury
Brief Title: Effects of Transcranial Direct Current Stimulation (tDCS) and Visual Illusion on Chronic Pain Due to Spinal Cord Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties and stopped funding
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Felipe Fregni, Principal Investigator, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010-p-001978
Record Dates: First submitted 2011-06-29; First posted 2011-07-27 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Chronic Pain; Spinal Cord Injury
Keywords: transcranial direct current stimulation
MeSH Terms: conditions — Chronic Pain; Spinal Cord Injuries | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (3):
- Active tDCS + visual illusion (Experimental): Subjects will receive active tDCS while watching a visual illusion movie (legs walking on a treadmill). Stimulation will last for 20 minutes.
  Interventions: Procedure: Transcranial Direct Current Stimulation (tDCS)
- Sham tDCS + visual illusion (Sham Comparator): Subjects will receive sham tDCS stimulation (30 seconds ramp up/ramp down) while watching a visual illusion movie (legs walking on a treadmill)
  Interventions: Procedure: Transcranial Direct Current Stimulation (tDCS)
- Healthy Subjects (Other): Healthy subjects will receive both interventions (active and sham) in a randomized and counterbalanced order. Each stimulation session will be at least 1 week apart to prevent carry-over effects
  Interventions: Procedure: Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Procedure: Transcranial Direct Current Stimulation (tDCS) — Subjects will undergo tDCS stimulation. For both active and sham stimulation, we will use electrodes of 35cm^2, at an intensity of 2mA. For active tDCS, the subject will undergo stimulation for 20 minutes. For sham stimulation, the current will be ramped up and then down again (for 30 seconds total) to simulate the feeling of active stimulation.
  Other Names: low intensity 1x1 direct current stimulator

SUMMARY:
The purpose of this study is to investigate the effects of Transcranial Direct Current Stimulation (tDCS) combined with watching a visual illusion on chronic pain due to spinal cord injury. The investigators hypothesize that active tDCS will reduce pain in subjects with spinal cord injury when compared to sham stimulation. The investigators will also measure changes in EEG data (alpha and beta frequencies) as well as motor cortex excitability.

ELIGIBILITY:
STUDY ELIGIBILITY CRITERIA

Inclusion Criteria:

1. Providing informed consent to participate in the study
2. 18 to 64 years old
3. With traumatic spinal cord injury (complete or incomplete) - for instance, due to fall, car accident or gun shot; (for spinal cord injury only)
4. Stable chronic pain for at least the three preceding months (for spinal cord injury only)
5. Score higher or equal to 4cm (0 cm= 'no pain' and 10cm='worst possible pain') on the Visual Analogue Scale (VAS) for pain perception at the baseline/start of the treatment (for spinal cord injury only)
6. Refractoriness to drugs for pain relief - such as tricyclic antidepressants, antiepileptic drugs and/or narcotics (pain resistant to at least 2 of these drugs supplied in adequate dosages for six months) (for spinal cord injury only)
7. Pain is not attributable to other causes, such as peripheral inflammation

Exclusion Criteria:

1. Clinically significant or unstable medical or psychiatric disorder
2. History of substance abuse
3. Neuropsychiatric comorbidities, including: Documented traumatic brain injury (TBI), defined as damage to brain tissue caused by an external mechanical force as evidenced by: loss of consciousness due to brain trauma, or post traumatic amnesia (PTA), or skull fracture, or objective neurological findings that can be reasonably attributed to TBI as assessed by the study PI
4. Implanted devices for pain control, such as vagal or deep brain stimulators
5. Contraindications to tDCS:

   * metal in the head
   * implanted brain medical devices
6. Pregnancy
7. Use of ventilators or ventilation support
8. Complete tetraplegic lesion (no motor function in the arms) (C3 to C8) as we will be measuring the motor evoked potential in the FDI (upper limbs); only tetraplegic patients with incomplete functional status and also as defined by the ability to elicit MEP in the FDI will be able to participate in this study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2010-12; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Changes in EEG (alpha and beta activity) | Measured for approximately 6 weeks
  Determine whether treatment with tDCS coupled with visual illusion change cortical activity as assessed with electroencephalography (EEG). We hypothesize that tDCS plus visual illusion increase in alpha activity and inhibit beta activity and this will be associated with pain reduction in patients with moderate to severe below-level spinal cord injury (SCI) pain. EEG measurements will take place throughout the subject's participation in the study, measured at: baseline, immediately pre- and post- stimulation and at follow-up visits for a total of approximately 6 weeks.

SECONDARY OUTCOMES:
Changes in cortical excitability | Measured for approximately 6 weeks
  To investigate whether active tDCS combined with visual illusion induces changes in motor cortex and as indexed by single and paired-pulse transcranial magnetic stimulation (TMS) as compared with sham tDCS coupled with visual illusion. We will also determine whether these changes are correlated with the clinical outcome (pain reduction). TMS measurements will take place throughout the subject's participation in the study, measured at: baseline, immediately pre- and post- stimulation and at follow-up visits for a total of approximately 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Fregni, MD, PhD, MPH, Principal Investigator — Spaulding Rehabilitation Hospital (SRH)
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States